CLINICAL TRIAL: NCT02035319
Title: Effect of Laser Treatment on Capillary Malformations Using Skin Imaging and Analysis
Brief Title: Effect of Laser Treatment on Capillary Malformations
Status: Withdrawn | Type: Observational
Why Stopped: No enrollments
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: Laser Capillary Malformation
Record Dates: First submitted 2014-01-07; First posted 2014-01-14 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Capillary Malformation; Port Wine Stain
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Port-Wine Stain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- capillary malformation treated by laser: capillary malformation treated by laser

SUMMARY:
In this research study investigators want to learn more about capillary malformations which are also known as port wine stains.

Investigators are asking children with capillary malformations (port wine stains) to be in the research, because investigators do not have a good idea of what to expect from the current treatments of these malformations. These malformations are treated with laser as clinically indicated and there are no standardized methods to assess improvement.

DETAILED DESCRIPTION:
Capillary malformations, specifically port wine stains, occur in one of every 12,000 live births (0.3% of newborns) with 90% on the face or neck. Pulsed dye laser therapy targeted at hemoglobin (i.e., 585 nm ± 5 nm) is commonly used to lessen the visual coloration and increase skin lightness. Presently, the outcomes of laser treatment are difficult to predict, in part due to the difficulty in quantifying the tissue changes with visual inspection methods. Quantitative skin imaging methods are currently being applied to measure the features and response to treatment for infantile hemangiomas. The current study proposes to apply these methods in the treatment of capillary malformations, e.g., port wine stains. The purpose is to determine (1) the effects of laser treatment on capillary malformations (using quantitative skin imaging methods and standard clinical assessment and (2) the relationships between the imaging outcomes immediately after treatment and after healing. In the within-subject design we aim to measure color, temperature, blood concentration and tissue mechanical properties for the capillary malformation relative to an un-involved site at baseline (prior to treatment), immediately following laser surgery and over time. Imaging outputs will be compared to the standard clinical evaluation in up to 100 patients from the Hemangioma and Vascular Malformation Center (HVMC) at regular intervals to determine changes over time. Skin sites will be imaged for color (size, erythema, blue color, lightness, excess erythema, uniformity), thermography, blood concentration and tissue mechanical properties (e.g., elasticity). Skin characteristics will be examined at baseline, prior to surgery, immediately following laser treatment, just prior to discharge and at 2 and 4-6 weeks following treatment. For subjects receiving multiple laser treatments, the procedures will be repeated after each surgery. Enrollment will occur over 2 years. Patients will be evaluated for a period of up to 6 months following the last surgery. We expect the research to provide objective measures to clarify the effectiveness of laser treatment and permit effective measurement of tumor response for therapeutic protocols.

ELIGIBILITY:
Inclusion Criteria:

* age 0-17
* Diagnosis of a capillary malformation
* Scheduled to undergo laser treatment of the capillary malformation
* Able to tolerate imaging procedures

Exclusion Criteria:

* Not scheduled to undergo laser treatment for capillary malformation
* Other vascular anomaly
* Not able to tolerate imaging procedures

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The research will be conducted among up to 100 patients of the Hemangioma and Vascular Malformation Center at Cincinnati Children's Hospital Medical Center who will undergo laser treatment for capillary malformations.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in capillary malformations in response to laser treatment | an expected average of 6 months
  Skin sites will be imaged for color (size, erythema, blue color, lightness, excess erythema, uniformity), thermography, blood concentration and tissue mechanical properties (e.g., elasticity).

SECONDARY OUTCOMES:
Number of patients with improvement in standard clinical evaluations compared to improvement as seen by quantitative imaging techniques in capillary malformations after laser treatment | an expected average of 6 months
  clinical characteristics of color clinical characteristics of temperature clinical characteristics of tissue morphology clinical characteristics of pliability clinical characteristics of hyperplasia digital imaging for color digital image processing thermal imaging image co-registration blood concentration biomechanical properties
Change in imaging outcome measures | an expected average of 6 months
  digital imaging for color digital image processing thermal imaging image co-registration blood concentration biomechanical properties

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Hammill, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States